CLINICAL TRIAL: NCT02452151
Title: Santeon InflixMab biosimILAr Research A Randomized, Controlled, Double Blind, Phase 4 Noninferiority Trial to Assess Efficacy of Infliximab-biosimilar (Inflectra) Compared to Infliximab-innovator (Remicade) in Patients With Inflammatory Bowel Disease in Remission.
Brief Title: "Efficacy and Safety of Infliximab-biosimilar (Inflectra) Compared to Infliximab-innovator (Remicade) in Patients With Inflammatory Bowel Disease in Remission: the SIMILAR Trial"
Acronym: SIMILAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Santeon (Unknown)
Responsible Party: Principal Investigator, J.M. Jansen, MD, J.M. Jansen, MD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIMILAR
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Colitis, Ulcerative; Crohn's Disease
Keywords: Inflectra; Infliximab; Biosimilar
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab-biosimilar (Experimental): Infliximab-Biosimilar (Inflectra) (5mg/kg or 10mg/kg) by intravenous (IV) infusion administered as a 2-hour infusion per dose as treatment. In total 4 to 6 doses of the study drug will be administered while continuing patient's dosing intervals, ranging between 6 to 10 weeks.
  Interventions: Drug: Infliximab-Biosimilar
- Infliximab-Innovator (Active Comparator): Infliximab-Innovator (Remicade) (5mg/kg or 10mg/kg) by intravenous (IV) infusion administered as a 2-hour infusion per dose as treatment. In total 4 to 6 doses of the study drug will be administered while continuing patient's dosing intervals, ranging between 6 to 10 weeks.
  Interventions: Drug: Infliximab-Innovator

INTERVENTIONS:
Drug: Infliximab-Biosimilar
  Arms: Infliximab-biosimilar
Drug: Infliximab-Innovator
  Arms: Infliximab-Innovator

SUMMARY:
The objective of this study is to compare the efficacy of Infliximab-Biosimilar to Infliximab-Innovator and to demonstrate its noninferiority, in patients with ulcerative colitis or Crohn's disease in remission under treatment with infliximab up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patients, male or female, aged above 18 years at time of enrolment will be selected from hospital databases based on appointments for Infliximab infusion as treatment for IBD. Patients are eligible for inclusion if they have an established diagnosis of ulcerative colitis or Crohn's disease, are in clinical remission and are medically treated with Infliximab for at least 12 weeks prior to inclusion.

Exclusion Criteria:

1. Patient has an allergy or hypersensitivity to one of the components of infliximab and/or immunoglobulin products, except hypersensitivity reactions which have a positive response to hydrocortisone and thereby are under control.
2. Patient has a current diagnosis with hepatitis B, hepatitis C or an infection with human immunodeficiency virus (HIV)-1 or 2. Patients with a past history of chronic hepatitis B or hepatitis C will not be excluded.
3. Patient has a history of tuberculosis (TB) or a current diagnosis of TB or other severe or chronic infection such as abscess, opportunistic infection or invasive fungal infection. Patients with a past history of a severe or chronic infection will not be excluded.
4. Patient has had recent exposure to persons with active TB. In that case screening for latent TB (defined as a positive result for interferon-γ release assay (IGRA) with a negative examination of chest X-ray) will be performed. If there is sufficient documentation of prophylaxis or complete resolution following TB-treatment based on hospital-specific guidelines the patient can be enrolled. If the result of the IGRA is indeterminate at screening, 1 retest will be done. If the repeated IGRA result is indeterminate again, the patient will be excluded. Patients with a positive IGRA result and a negative examination of chest X-ray who has received at least the first 30 days of TB-therapy can be enrolled.
5. Patient who is taking any of the following concomitant medications or treatment:

   * Corticosteroids (prednisone, prednisolone or budosenide).
   * Live or live-attenuated vaccine within 8 weeks of randomization.
   * Any other biological treatments than infliximab.
   * Subtotal and total colectomy prior to randomization.
   * Any planned abdominal surgery for IBD at the time of randomization and/or during the study period.
6. Patient has one or more of the following medical conditions:

   * Active entero-vesical, entero-retroperitoneal, entero-cutaneous and entero-vaginal fistula for within 6 months prior to screening. Entero-enteral fistulae without clinical significant symptoms upon investigator's opinion and anal fistulae without draining problems are allowed.
   * Current short bowel syndrome.
   * History of any malignancy within the 5 years prior to randomization except cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma or completely excised and cured squamous carcinoma of the uterine cervix.
   * History of lymphoma or lymphproliferative disease or bone marrow hyperplasia.
   * New York Heart Association (NYHA) class III or IV heart failure.
   * History of organ transplantation, including corneal graft/transplantation.
7. Patient has had treatment with any other investigational device or medical product within 4 weeks of randomization or 5 half-lives, whichever is longer.
8. Female patient who is currently pregnant, breastfeeding or planning to become pregnant or breastfeed within 6 months of the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 3 months
  Efficacy of Infliximab-Biosimilar and Infliximab will be assessed by evaluation of the relapse rate for each diagnosis seperately.
Duration of clinical remission | 3 months
  Efficacy of Infliximab-Biosimilar and Infliximab will be assessed by evaluation of the the duration of clinical remission for each diagnosis seperately.